CLINICAL TRIAL: NCT04826146
Title: Monitoring the Depth of Anesthesia Using the qCON and qNOX Indices During Pediatric Surgery: a Multi-centre Study
Brief Title: Pediatric Validation of CONOX Monitor During Surgery
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Patricio Gonzalez Pizarro (Other)
Responsible Party: Sponsor-Investigator, Patricio Gonzalez Pizarro, Principal Investigator, Hospital Universitario La Paz
Organization: Hospital Universitario La Paz (Other)
Other Study IDs: PI-3871
Record Dates: First submitted 2021-03-21; First posted 2021-04-01 (Actual); Last update posted 2021-09-09 (Actual); Status verified 2021-09

CONDITIONS: Anesthesia; Anesthesia Awareness; Nociceptive Pain; Pediatric ALL; Surgery; Pain
MeSH Terms: conditions — Intraoperative Awareness; Nociceptive Pain; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- CONOX: Patients are monitored with BIS and CONOX
  Interventions: Device: Validation of qCON versus BIS

INTERVENTIONS:
Device: Validation of qCON versus BIS — Correlation between qCON and BIS values (main outcome) and qNOX and MOAA/S scale are determined
  Other Names: Validation of qNOX Vs MOAA/S Scale

SUMMARY:
Pediatric Validation of CONOX Monitoring device (qCON and qNOX indices) for anesthesia depth during surgery

ELIGIBILITY:
Inclusion Criteria:

* General Anesthesia using propofol, sevoflurane or desflurane
* ASA I - IV
* Surgical procedure longer than 60 minutes

Exclusion Criteria:

* Neurological disorders
* Inability to correctly place BIS and CONOX probes in forehead
* Pregnancy
* Active prescription for drugs involving chronic pain and / or central nervous system
* Hemodynamic instability

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Children undergoing general anesthesia for a surgical procedure longer than 60 minutes
Sampling Method: Non-Probability Sample
Enrollment: 65 (Estimated)
Dates: Start 2020-07-01 (Actual); Primary Completion 2021-12-01 (Estimated); Study Completion 2021-12-30 (Estimated)

PRIMARY OUTCOMES:
Correlation of qCOX and BIS values | prospective data acquisition through study completion, an average of 1 year
  Both values are correlated by a blind investigator

SECONDARY OUTCOMES:
Correlation of qNOX and MOAA/S values | prospective data acquisition through study completion, an average of 1 year
  Both values are correlated by a blind investigator

CONTACTS AND LOCATIONS:
Locations (2):
- Spain (2):
  - Hospital Universitario La Paz, Madrid
  - Hospital Universitario de Santiago de Compostela (CHUS), Santiago de Compostela

IPD SHARING:
Plan to Share IPD: Undecided